CLINICAL TRIAL: NCT00006355
Title: Phase I/II Study of Pyrazoloacridine (PZA) in Adults With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Pyrazoloacridine Followed by Radiation Therapy in Treating Adults With Newly Diagnosed Supratentorial Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTT-9804 CDR0000068223; U01CA062475 (NIH); P30CA006973 (NIH); NABTT-9804; JHOC-NABTT-9804
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — NSC 366140; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: pyrazoloacridine
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of pyrazoloacridine followed by radiation therapy in treating adults who have newly diagnosed supratentorial glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose, toxicity, and pharmacokinetics of pyrazoloacridine in adults with newly diagnosed, supratentorial glioblastoma multiforme treated with pyrazoloacridine followed by radiotherapy.
* Determine the response rate, duration of disease free survival, and survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to type of anticonvulsant (hepatic metabolic enzyme inducers vs hepatic metabolic enzyme moderate inducers or noninducers).

Patients receive pyrazoloacridine (PZA) IV over 3 hours on day 1. Treatment repeats every 3 weeks for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity. Following completion of PZA treatment, patients undergo cranial irradiation 5 days a week for 6 weeks.

Cohorts of 3 patients receive escalating doses of PZA until the maximum tolerated dose (MTD) is determined. Additional patients receive PZA at the MTD.

Patients are followed monthly for survival.

PROJECTED ACCRUAL: A minimum of 3 patients will be accrued for phase I and a total of 18-35 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven, newly diagnosed, supratentorial, grade IV astrocytoma (glioblastoma multiforme)

  * Incompletely resected disease
* Must have measurable and contrast enhancing tumor on the postoperative MRI/CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.7 mg/dL

Other:

* No other serious concurrent infection or medical illness that would preclude study therapy
* No other active malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer
* No psychosis requiring ongoing therapy with antipsychotic medication
* Mini mental score at least 15
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy or biologic agents (including immunotoxins, immunoconjugates, antisense compounds, peptide receptor antagonists, interferons, interleukins, tumor infiltrating lymphocytes, lymphokine activated killer cells, or gene therapy) for glioblastoma multiforme
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy:

* No prior chemotherapy for glioblastoma multiforme

Endocrine therapy:

* No prior hormonal therapy for glioblastoma multiforme
* Prior glucocorticoids allowed
* Concurrent corticosteroids allowed if on stable dose (no increase within the past 5 days)

Radiotherapy:

* No prior radiotherapy for glioblastoma multiforme

Surgery:

* See Disease Characteristics
* Recovered from immediate postoperative period

Other:

* Greater than 10 days since prior anticonvulsants that induce hepatic metabolic enzymes (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or felbamate)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05; Primary Completion 2004-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (8):
- United States (8):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Frenay M, Lebrun C, Fontaine D, et al.: First-line chemotherapy in non resectable low-grade astrocytomas in adults. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2095, 71b, 2002.
- [Result] Lesser GJ, Carson K, Supko J, et al.: A phase I/II trial and pharmacokinetic study of pyrazoloacridine in adults with newly diagnosed glioblastoma multiforme. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-485, 121a, 2003.
- [Result] Lesser GJ, Carson K, Priet R, et al.: A phase I/II trial of pyrazoloacridine (PZA) in adults with newly diagnosed glioblastoma multiforme (GBM). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2097, 2002.